CLINICAL TRIAL: NCT06864234
Title: Effect of Beta-blockers on Coronary Flow and Resistance in Patients With ANOCA: a Randomised, Placebo-controlled, Mechanistic Study
Brief Title: Effect of Beta-blockers on Coronary Flow and Resistance in Patients With ANOCA
Acronym: BEACON
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VZW Cardiovascular Research Center Aalst (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2025/032
Record Dates: First submitted 2025-03-02; First posted 2025-03-07 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Coronary Arterial Disease (CAD); Angina (Stable); Microvascular Circulation
Keywords: angina; coronary artery disease; absolute coronary flow; continuous intracoronary thermodilution; Beta-blockers
MeSH Terms: conditions — Angina, Stable; Angina Pectoris; Coronary Artery Disease | interventions — Sodium Chloride; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): IV 0.9% NaCl (5 ml)
  Interventions: Drug: Saline (NaCl)
- Beta-blocker (Active Comparator): IV metoprolol (5 ml of 1 mg/ml solution for injection)
  Interventions: Drug: Metoprolol Tartrate

INTERVENTIONS:
Drug: Saline (NaCl) — IV 0.9% NaCl (5 ml)
  Arms: Placebo
Drug: Metoprolol Tartrate — Metoprolol Tartrate (5 ml of 1 mg/ml solution for injection)
  Arms: Beta-blocker

SUMMARY:
The goal of this clinical trial is to learn whether beta-blockers can improve coronary blood flow and reduce resistance in patients with angina and no obstructive coronary arteries (ANOCA).

The main questions it aims to answer are:

* Do beta-blockers improve coronary blood flow in patients with ANOCA?
* Do beta-blockers reduce coronary microvascular resistance in these patients?

Researchers will compare a beta-blocker to a placebo to see if the medication has measurable effects on coronary circulation.

Participants will:

* Receive a beta-blocker or a placebo
* Undergo specialized heart tests (such as coronary flow and resistance measurements) before and after treatment.

DETAILED DESCRIPTION:
INTRODUCTION

Beta-blockers (BB) remain a mainstay in the management of cardiac diseases due to a wide range of cardiovascular effects. Through the antagonism of beta-adrenergic stimuli, BB reduce heart rate, cardiac contractility, and left ventricular wall stress, with the latter mediated in part by the antihypertensive action of the drug class. Whilst first-generation BB, such as propranolol, block both β1 and β2 adrenoceptors, second-generation BB (e.g. metoprolol and atenolol) are selective for β1 adrenoceptors and thus avoid the side effects seen with unwanted β2 adrenoceptor blockade, making them ideal antianginal and antiarrhythmic drugs. Third-generation BB - namely carvedilol and nebivolol - exert an additional vasodilatory effect through α-adrenoreceptor blockade and increased nitric oxide (NO) production, respectively, making them effective choices in the management of heart failure and hypertension.

Most recently, BB have been recommended for the treatment of coronary microvascular dysfunction (CMD). CMD is an increasingly recognised pathology affecting patients both with and without coronary artery disease. Its treatment with drugs such as BB has been shown to improve both symptoms and quality of life, leading to its inclusion in the latest European and American guidelines.

Yet, whilst numerous studies have assessed the cardiovascular effects of beta-blockers, many have yielded discordant results regarding their effect on coronary function. Billinger et al. found that IV metoprolol was associated with a significant increase in hyperaemic flow as measured by intracoronary Doppler, with a corresponding decrease in total coronary resistance, among patients with epicardial disease. However, a later study by Togni et al. employing intracoronary Doppler before and after the administration of intracoronary nebivolol, reported a significant increase in coronary flow reserve (CFR) driven by a reduction in resting flow in patients without CAD, and an increase in maximal coronary flow in patients with CAD.

Studies employing nuclear imaging have also yielded inconsistent results. Böttcher et al. found that healthy volunteers who underwent 13N-ammonia PET at baseline and 1 hour after the administration of 50 mg of oral metoprolol exhibited a decrease in resting myocardial blood flow (MBF) in line with a corresponding decrease in cardiac work, but a significant increase in hyperaemic MBF. This ultimately resulted in an increase in CFR. Conversely, Koepfli et al. reported a significant decrease in resting myocardial blood flow but no significant change in hyperaemic MBF in 36 CAD patients who underwent 13N-ammonia PET before and after 12 weeks of oral metoprolol or carvedilol. Studies employing transthoracic Doppler have also reported discordant results.

Beyond the discordant results produced by many of these studies, there are several limitations associated with this work. First, no studies have employed a strict randomised, placebo-controlled design to isolate the true coronary effects of beta-blockers. Second, no studies have specifically explored the effect of BB on patients with ANOCA or CMD, an increasingly recognised patient group for which BB represent a guideline-recommended treatment. Third, there have been no studies that have specifically assessed the effect of BB on coronary microvascular function; by focusing on flow and CFR, a global coronary index that is not specific to the microvascular compartment, previous work has only assessed the effect of BB on overall coronary function without isolating their effect on the epicardial or microvascular compartments. Finally, none of these studies have employed continuous intracoronary thermodilution, a novel assessment modality that permits the precise and accurate measurement of absolute coronary flow and resistance in humans. This extensively validated technique permits the detailed assessment of the epicardial and microvascular compartments in isolation and has opened the door to previously inaccessible physiological studies.

GOAL OF THE STUDY

In the present study, continuous intracoronary thermodilution will be used to assess the cardiovascular effects of intravenous BB compared with a placebo control, with a focus on metrics of microvascular function, such as microvascular resistance and microvascular resistance reserve (MRR).

DESIGN

This is an investigator-initiated, prospective, double-blinded, randomised controlled study recruiting patients from a single centre undergoing diagnostic coronary angiography who are found to have angina and non-obstructive coronary arteries (ANOCA). Patients will be randomised between intravenous BB and placebo.

OVERVIEW OF THE STUDY PROTOCOL

Given that this is a mechanistic trial aiming to elucidate the true cardiovascular effects of BB, all recruited patients will have any pre-existing BB therapy/other vasoactive medications stopped 24 hours before the protocol.

(i) Protocol

The following protocol will be performed:

1. Diagnostic angiography: ensure no vasodilatory medications are given e.g. nicardipine or nitrates
2. Baseline left ventricular end-diastolic pressure (LVEDP): obtained using a standard pigtail catheter. Left ventricular angiography will not be performed.
3. Baseline continuous intracoronary thermodilution: performed to obtain both resting and hyperaemic pressure (Pd and Pa), volumetric blood flow (Q), and resistance measurements (R). These measurements require the use of a pressure/temperature guidewire and a dedicated infusion catheter. They are performed routinely in our clinical practice to evaluate microvascular function. The continuous intracoronary thermodilution technique is described in detail below (see paragraph 'Continuous thermodilution measurements').
4. Randomisation: following the measurement of baseline resting and hyperaemic values, the patient will be randomised to either IV metoprolol or placebo (IV 0.9% NaCl of equivalent volume) by the research nurse. The research nurse will administer the intervention with both physicians and the patient blinded to patient randomisation.
5. Repeat continuous intracoronary thermodilution: the same resting and hyperaemic measurements will be repeated 10 minutes after the administration of the intervention.

It is expected that the protocol, including the recording of both baseline and post-intervention values, will last ~15 minutes.

(ii) Randomisation Randomisation will be performed using the concealed envelope system by a dedicated study nurse in line with the pre-specified sample size calculation. Patients, operators, and all other clinical team members will be blinded to randomisation.

(iii) Measured parameters The following parameters will be recorded/calculated for rest and hyperaemic at both baseline as well as at 10 minutes after the administration of the intervention to capture the full effect of BB on both coronary and systemic haemodynamics.

* Absolute coronary blood flow (Q)
* Microvascular resistance (Rµ)
* Epicardial resistance (Repi)
* Total resistance (Rtot)
* Aortic pressure (Pa)
* Distal coronary pressure (Pd)
* Coronary flow reserve (CFR)
* Microvascular resistance reserve (MRR)
* Systolic pressure-time index (SPTI) i.e. area under the Pa curve.
* Buckberg index (estimate of myocardial perfusion) i.e. diastolic pressure-time index (i.e. time of coronary perfusion) divided by systolic pressure-time index (i.e. time of myocardial oxygen demand).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing diagnostic coronary angiography for suspected angina pectoris who are found to have ANOCA i.e. an FFR >0.80 and no diameter stenosis >50%
* Normal, TIMI 3 flow at angiography
* Stable haemodynamics

Exclusion Criteria:

* Clinical signs or symptoms of congestive heart failure
* Severe valvular heart disease requiring either surgical or percutaneous intervention
* History of coronary artery bypass grafting
* Tortuous coronary anatomy in which wire manipulation could be complex
* Heart rate <60 beats per minute
* Systolic blood pressure <100 mmHg
* Unable to give consent
* LVEF<40%

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the absolute coronary flow 10 minutes after administration of the intervention | 10 minutes from the administration of the intervention
  Absolute coronary flow will be measured using continuous intracoronary thermodilution
Change from baseline in the absolute microvascular resistance 10 minutes after administration of the intervention | 10 minutes from the administration of the intervention
  Absolute microvascular resistance will be calculated using absolute coronary flow and distal coronary pressure
Change from baseline in the microvascular resistance reserve (MRR) 10 minutes after administration of the intervention | 10 minutes from the administration of the intervention
  MRR will be calculated using absolute coronary flow, aortic pressure and distal coronary pressure

SECONDARY OUTCOMES:
Change from baseline in the coronary flow reserve (CFR) 10 minutes after administration of the intervention | 10 minutes from the administration of the intervention
  CFR will be calculated using absolute coronary flow
Change from baseline in the absolute epicardial resistance 10 minutes after administration of the intervention | 10 minutes from the administration of the intervention
  Absolute epicardial resistance will be calculated using absolute coronary flow, aortic pressure and distal coronary pressure
Change from baseline in aortic pressure 10 minutes after administration of the intervention | 10 minutes from the administration of the intervention
  Aortic pressure will be measured using the coronary guiding catheter
Change from baseline in distal coronary pressure 10 minutes after administration of the intervention | 10 minutes from the administration of the intervention
  Distal coronary pressure will be measured using a standard coronary pressure wire
Change from baseline in left ventricular end-diastolic pressure 10 minutes after administration of the intervention | 10 minutes from the administration of the intervention
  LVEDP will be measured using a pigtail catheter at baseline, and at the end of the protocol
Change from baseline in left ventricular work 10 minutes after administration of the intervention | 10 minutes from the administration of the intervention
  Left ventricular work will be estimated using the systolic pressure-time index (SPTI) derived from the aortic pressure curve.
Change from baseline in myocardial perfusion 10 minutes after administration of the intervention | 10 minutes from the administration of the intervention
  Myocardial perfusion will be estimated using the Buckberg Index. It will be calculated by dividing the diastolic pressure-time index (i.e. time of coronary perfusion) by the systolic pressure-time index (i.e. time of myocardial oxygen demand).

CONTACTS AND LOCATIONS:
Locations (1):
- OLV Cardiovascular Center Aalst, Aalst, Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No
This was included in the original ethical committee sumission

REFERENCES:
- [Background] Erdogan D, Gullu H, Caliskan M, Ciftci O, Baycan S, Yildirir A, Muderrisoglu H. Nebivolol improves coronary flow reserve in patients with idiopathic dilated cardiomyopathy. Heart. 2007 Mar;93(3):319-24. doi: 10.1136/hrt.2006.091751. Epub 2006 Oct 25. PMID 17065184
- [Background] Galderisi M, Cicala S, D'Errico A, de Divitiis O, de Simone G. Nebivolol improves coronary flow reserve in hypertensive patients without coronary heart disease. J Hypertens. 2004 Nov;22(11):2201-8. doi: 10.1097/00004872-200411000-00024. PMID 15480106
- [Background] Koepfli P, Wyss CA, Namdar M, Klainguti M, von Schulthess GK, Luscher TF, Kaufmann PA. Beta-adrenergic blockade and myocardial perfusion in coronary artery disease: differential effects in stenotic versus remote myocardial segments. J Nucl Med. 2004 Oct;45(10):1626-31. PMID 15471825
- [Background] Bottcher M, Czernin J, Sun K, Phelps ME, Schelbert HR. Effect of beta 1 adrenergic receptor blockade on myocardial blood flow and vasodilatory capacity. J Nucl Med. 1997 Mar;38(3):442-6. PMID 9074535
- [Background] Togni M, Vigorito F, Windecker S, Abrecht L, Wenaweser P, Cook S, Billinger M, Meier B, Hess OM. Does the beta-blocker nebivolol increase coronary flow reserve? Cardiovasc Drugs Ther. 2007 Apr;21(2):99-108. doi: 10.1007/s10557-006-0494-7. PMID 17235472
- [Background] Billinger M, Seiler C, Fleisch M, Eberli FR, Meier B, Hess OM. Do beta-adrenergic blocking agents increase coronary flow reserve? J Am Coll Cardiol. 2001 Dec;38(7):1866-71. doi: 10.1016/s0735-1097(01)01664-3. PMID 11738286